CLINICAL TRIAL: NCT02680977
Title: Mucuna Pruriens Therapy in Parkinson's Disease: a Double-blind, Placebo-controlled, Randomized, Crossover Study.
Brief Title: Mucuna Pruriens Therapy in Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ASST Gaetano Pini-CTO (Other)
Collaborators: Grisons Foundation for Parkinson's Disease (Other)
Responsible Party: Principal Investigator, Roberto Cilia, Neurologist, ASST Gaetano Pini-CTO
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBN.SC.013/2015
Record Dates: First submitted 2016-02-09; First posted 2016-02-12 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Parkinson's Disease
Keywords: Mucuna pruriens; Levodopa
MeSH Terms: conditions — Parkinson Disease | interventions — Benserazide; benserazide, levodopa drug combination; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- MP-Equivalent; MP-Low; MP+DDCI (Experimental): MP-Equivalent: Mucuna pruriens powder at equivalent dosage than LD+DDCI. The dose of MP is calculated to obtain a 5-fold Levodopa dose than LD+DDCI (for example 100mg of Madopar corresponds to 500mg of Levodopa in MP).
  MP-Low: Mucuna pruriens powder at low dosage. The dose of MP is calculated to obtain a 3.5-fold Levodopa content than LD+DDCI (for example 100mg of Madopar corresponds to 350mg of Levodopa in MP) MP+DDCI: Mucuna pruriens powder plus Benserazide. The dosage of MP is calculated to obtain the same Levodopa content than LD+DDCI (for example 100mg of Madopar corresponds to 100mg of Levodopa in MP plus 25mg of Benserazide)
  Interventions: Other: MP-Equivalent; Other: MP-Low; Other: MP+DDCI
- LD+DDCI; LD-DDCI (Active Comparator): LD+DDCI: Levodopa plus Benserazide (dispersible formulation). The dose is calculated as 3.5mg per kg of body weight.
  LD-DDCI: Levodopa without any dopa decarboxylase inhibitor (galenic formulation). The dose is 5-fold than LD+DDCI.
  Interventions: Drug: LD+DDCI; Drug: LD-DDCI
- Placebo (Placebo Comparator): Powder of groundnuts
  Interventions: Other: Placebo

INTERVENTIONS:
Other: MP-Equivalent — Mucuna pruriens powder at equivalent dosage than LD+DDCI. The dose of MP is calculated to obtain a 5-fold Levodopa dose than LD+DDCI.
  Other Names: Mucuna pruriens at equivalent dose than LD-DDCI
  Arms: MP-Equivalent; MP-Low; MP+DDCI
Other: MP-Low — Mucuna pruriens powder at low dosage. The dose of MP is calculated to obtain a 3.5-fold Levodopa content than LD+DDCI
  Other Names: Mucuna pruriens at low dosage
  Arms: MP-Equivalent; MP-Low; MP+DDCI
Other: MP+DDCI — Mucuna pruriens powder plus Benserazide. The dosage of MP is calculated to obtain the same Levodopa content than LD+DDCI. Benserazide is given as 1:4 ratio with Levodopa.
  Other Names: Mucuna pruriens plus Benserazide
  Arms: MP-Equivalent; MP-Low; MP+DDCI
Drug: LD+DDCI — Levodopa plus Benserazide
  Other Names: Madopar
  Arms: LD+DDCI; LD-DDCI
Drug: LD-DDCI — Levodopa without any DDCI
  Other Names: Levodopa without any DDCI (galenic formulation)
  Arms: LD+DDCI; LD-DDCI
Other: Placebo — Groundnuts powder
  Arms: Placebo

SUMMARY:
In low-income areas worldwide, most patients with Parkinson's disease (PD) cannot afford long-term Levodopa therapy. A potential therapeutic option for them is the use of a legume called Mucuna Pruriens var. Utilis (MP), which has seeds with a high levodopa content (5-6%) and grows in all tropical areas of the world. MP powder is very cheap (total annual cost for a PD patient: 10-15 US $). The aim of this study is to assess efficacy and tolerability of acute and chronic use of MP compared to standard Levodopa therapy.

The primary objective of this study is to investigate efficacy of acute levodopa challenge using MP in comparison to levodopa with a Dopa Decarboxylase Inhibitor (LD+DDCI) and without (LD-DDCI) and placebo.

The secondary objectives are to investigate safety of acute intake of MP as well as efficacy and safety of chronic intake of MP over a 8-week period in comparison to usual LD+DDCI home therapy.

DETAILED DESCRIPTION:
Background: Levodopa is the gold standard in the treatment of Parkinson's disease (PD). However, in low-income areas worldwide, most patients with PD cannot afford chronic therapy with levodopa. It is therefore mandatory to identify an interventional strategy designed to ease the economic burden of pharmacological management of PD in developing countries. A potential therapeutic option for them is the use of a legume called Mucuna Pruriens variant Utilis (MP), which has seeds containing high LD concentrations and grows spontaneously in all tropical and subtropical areas of the world, including South America, Africa and Asia. It is considered an invasive plant, as it grows rapidly without any particular measure needed to ensure its growth. The cost of home preparation of MP roasted powder is negligible and it is easy to store for a long time. LD was isolated from MP seeds for the first time in 1937 and its concentration therein was estimated to be 4-6%. MP is also known as Ayurvedic remedy for PD since ancient times.

Preliminary data: Published studies in parkinsonian rats, primates and humans suggest that MP may be used to improve PD motor symptoms without major side effects.

In a preliminary study, we analyzed 25 samples of MP from Africa, Latin America and Asia and measured the content in LD and anti-nutrients. We found that LD concentration in roasted powder samples was consistent with previous literature (median[Inter-Quartile Range] 5.3%[5.17-5.5]) and found no harmful anti-nutrients in all MP samples.

Study population: patients with diagnosis of idiopathic PD, including sustained response to levodopa and presence of motor fluctuations defined as predictable wearing-off, unpredictable ON-OFF fluctuations and sudden OFF periods.

Setting: Clinica Niño Jesus, Santa Cruz (Bolivia). This setting is chosen because the local neurologist Dr. Janeth Laguna has long-term experience on MP therapy in patients with PD (approximately 10 years). She started using MP because patients living in rural areas asked her to use this cheap source of LD to reduce the monthly cost of anti-PD therapy. In her experience, J.L. never recorded any serious adverse event (personal communication).

Preliminary Laboratory Test: The levodopa content in the powder obtained from roasted seeds of Bolivian black ecotype of MP was tested in a laboratory in Milan (Italy) and found to be 5.7%. No alkaloids or major antinutrients were found.

Objectives:

The primary objective is to assess the efficacy of acute challenge of MP roasted powder compared to Levodopa formulations with a dopa-decarboxylase inhibitor (LD-DDCI) and without (LD+DDCI), and placebo. Levodopa dose with DDCI is administered at 3.5 mg/kg, while Levodopa without DDCI is administered at the equivalent dose. This conversion factor is 5-fold, based on published studies comparing clinical and pharmacokinetic Levodopa effects with and without a DDCI and a previous double blind study on MP in patients with PD. For example, 100mg of Levodopa plus DDCI (either Benserazide or Carbidopa) corresponds to 500mg of Levodopa without any DDCI, obtained by administration of 8.75 grams of MP roasted powder (considering 5.7% of Levodopa in the bolivian ecotype of MP). Levodopa dose from MP is planned to be administered at not only at the equivalent dose of LD+DDCI (i.e. 5-fold), but also at the lower dosage of 3.5-fold.

Design: double-blind, randomized, placebo controlled, crossover study of acute response to levodopa-based therapies Duration: 3-6 hours for each treatment arm.

The secondary objectives include additional measures of efficacy of acute intake of MP as well as efficacy and safety of chronic use of MP as the only source of levodopa compared to optimized home LD+DDCI therapy. This latter part is performed after completion of the acute challenge part of the study.

Design: single-blind, randomized, crossover study of chronic response to levodopa-based therapies.

Duration: 8 weeks per treatment arm plus 3-week dose adjustment period. Initial levodopa-based therapy regimen (either MP therapy or Levodopa/Benserazide) may be adjusted for a period up to 3 weeks to optimize daily motor status during waking hours. After this period, patients enter the study and levodopa daily dose must be left unchanged throughout the 16-week course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic Parkinson's disease according to the United Kingdom Brain Bank criteria, defined by the presence of at least two of the cardinal signs of the disease (resting tremor, bradykinesia, rigidity) without any other known cause of parkinsonism.
* Sustained response to levodopa and presence of motor fluctuations for at least 1 h every day during waking hours, defined as predictable wearing-off, unpredictable ON-OFF fluctuations and sudden OFF periods.
* Patients had to receive optimum LD+DDCI, be stable for at least 30 days before baseline assessment.
* Availability to written informed consent

Exclusion Criteria:

* Cognitive impairment according to Mini-Mental State Examination < 26/30
* Clinically significant psychiatric illness, including psychosis, major depression and addiction disorders (including compulsive levodopa intake).
* Hoehn and Yahr stage of 5/5 in the medication-OFF state
* Severe, unstable medical conditions (i.e. unstable diabetes mellitus, moderate to severe renal or hepatic impairment, neoplasms)
* Risk of pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-02; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Magnitude of motor response | up to 3 hours
  Percentage of change in UPDRS motor score (part III) from baseline (overnight OFF state) to 90 minutes and 180 minutes after acute intake (full ON state)

SECONDARY OUTCOMES:
ON duration | up to 6 hours
  Duration of full ON state after acute intake
Latency to ON | up to 6 hours
  Latency in minutes between the acute intake (at the overnight OFF state) and the ON state
Severity of dyskinesias | up to 3 hours
  Severity of dyskinesias after acute intake, as assessed by the abnormal involuntary movements scale (AIMS) at 90 minutes and 180 minutes
Changes in vital signs | up to 3 hours
  Changes in blood pressure and heart rate at 90 minutes and 180 minutes after acute intake
Change in mean total daily off-time without troublesome dyskinesias | 16 weeks
  Change in mean total daily off-time as measured by 24-h diaries during chronic treatment
Change in quality of life questionnaire scores | 16 weeks
  Change in quality of life (as assessed by the PDQ-39) during chronic treatment
Change in Non-Motor Symptoms questionnaire scores | 16 weeks
  Change in non-motor symptoms (as assessed by the Movement Disorders Society - Non-Motor Symptoms questionnaire) during chronic treatment
Frequency of spontaneously reported adverse events | 16 weeks
  Incidence of spontaneously reported adverse events during acute and chronic treatment
Laboratory indices | 16 weeks
  Changes in laboratory indices from baseline to week 16
Electrocardiography | 16 weeks
  Changes in electrocardiographic measures from baseline to week 16

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Cilia, MD, Principal Investigator — ASST Gaetano Pini-CTO; Gianni Pezzoli, MD, Study Chair — ASST Gaetano Pini-CTO
Locations (1):
- Clinica Niño Jesus, Santa Cruz de la Sierra, Bolivia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Katzenschlager R, Evans A, Manson A, Patsalos PN, Ratnaraj N, Watt H, Timmermann L, Van der Giessen R, Lees AJ. Mucuna pruriens in Parkinson's disease: a double blind clinical and pharmacological study. J Neurol Neurosurg Psychiatry. 2004 Dec;75(12):1672-7. doi: 10.1136/jnnp.2003.028761. PMID 15548480
- [Background] Lieu CA, Kunselman AR, Manyam BV, Venkiteswaran K, Subramanian T. A water extract of Mucuna pruriens provides long-term amelioration of parkinsonism with reduced risk for dyskinesias. Parkinsonism Relat Disord. 2010 Aug;16(7):458-65. doi: 10.1016/j.parkreldis.2010.04.015. Epub 2010 May 31. PMID 20570206
- [Background] Contin M, Lopane G, Passini A, Poli F, Iannello C, Guarino M. Mucuna pruriens in Parkinson Disease: A Kinetic-Dynamic Comparison With Levodopa Standard Formulations. Clin Neuropharmacol. 2015 Sep-Oct;38(5):201-3. doi: 10.1097/WNF.0000000000000098. PMID 26366963
- [Background] Poddighe S, De Rose F, Marotta R, Ruffilli R, Fanti M, Secci PP, Mostallino MC, Setzu MD, Zuncheddu MA, Collu I, Solla P, Marrosu F, Kasture S, Acquas E, Liscia A. Mucuna pruriens (Velvet bean) rescues motor, olfactory, mitochondrial and synaptic impairment in PINK1B9 Drosophila melanogaster genetic model of Parkinson's disease. PLoS One. 2014 Oct 23;9(10):e110802. doi: 10.1371/journal.pone.0110802. eCollection 2014. PMID 25340511
- [Background] Lieu CA, Venkiteswaran K, Gilmour TP, Rao AN, Petticoffer AC, Gilbert EV, Deogaonkar M, Manyam BV, Subramanian T. The Antiparkinsonian and Antidyskinetic Mechanisms of Mucuna pruriens in the MPTP-Treated Nonhuman Primate. Evid Based Complement Alternat Med. 2012;2012:840247. doi: 10.1155/2012/840247. Epub 2012 Sep 10. PMID 22997535
- [Background] Bega D, Gonzalez-Latapi P, Zadikoff C, Simuni T. A review of the clinical evidence for complementary and alternative therapies in Parkinson's disease. Curr Treat Options Neurol. 2014 Oct;16(10):314. doi: 10.1007/s11940-014-0314-5. PMID 25143234
- [Background] Manyam BV. Paralysis agitans and levodopa in "Ayurveda": ancient Indian medical treatise. Mov Disord. 1990;5(1):47-8. doi: 10.1002/mds.870050112. PMID 2404203
- [Background] Behari M, Bhatnagar SP, Muthane U, Deo D. Experiences of Parkinson's disease in India. Lancet Neurol. 2002 Aug;1(4):258-62. doi: 10.1016/s1474-4422(02)00105-9. No abstract available. PMID 12849459
- [Background] Ovallath S, Deepa P. The history of parkinsonism: descriptions in ancient Indian medical literature. Mov Disord. 2013 May;28(5):566-8. doi: 10.1002/mds.25420. Epub 2013 Mar 8. PMID 23483637
- [Derived] Cilia R, Laguna J, Cassani E, Cereda E, Raspini B, Barichella M, Pezzoli G. Daily intake of Mucuna pruriens in advanced Parkinson's disease: A 16-week, noninferiority, randomized, crossover, pilot study. Parkinsonism Relat Disord. 2018 Apr;49:60-66. doi: 10.1016/j.parkreldis.2018.01.014. Epub 2018 Jan 11. PMID 29352722
- [Derived] Cilia R, Laguna J, Cassani E, Cereda E, Pozzi NG, Isaias IU, Contin M, Barichella M, Pezzoli G. Mucuna pruriens in Parkinson disease: A double-blind, randomized, controlled, crossover study. Neurology. 2017 Aug 1;89(5):432-438. doi: 10.1212/WNL.0000000000004175. Epub 2017 Jul 5. PMID 28679598
- Available data/document: Laboratory analysis (preliminary to clinical study) — http://www.mdsabstracts.com/abstract.asp?MeetingID=802&id=113641 — This study (currently submitted) describes the aims and results of laboratory testing on several different ecotypes of Mucuna pruriens, including the Bolivian variety to be used in the present protocol